CLINICAL TRIAL: NCT01555125
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Study of Subcutaneous Secukinumab in Prefilled Syringes to Demonstrate Efficacy After Twelve Weeks of Treatment, and to Assess the Safety, Tolerability, Usability and Long-term Efficacy in Subjects With Chronic Plaque-type Psoriasis
Brief Title: First Study of Secukinumab in Pre-filled Syringes in Subjects With Chronic Plaque-type Psoriasis: Response at 12 Weeks
Acronym: FEATURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2308; 2011-006057-28 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Moderate to Severe Plaque-type Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- secukinumab 150 mg (Experimental): Drug
  Interventions: Drug: secukinumab 150 mg
- secukinumab 300 mg (Experimental): Drug
  Interventions: Drug: secukinumab 300 mg
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: secukinumab 150 mg — After the data base lock of week 52 data has been performed, subjects will receive secukinumab 150 mg treatment as open label for the remainder of the extension treatment period
  Arms: secukinumab 150 mg
Drug: secukinumab 300 mg — After the data base lock of week 52 data has been performed, subjects will receive secukinumab 300 mg treatment as open label for the remainder of the extension treatment period
  Arms: secukinumab 300 mg
Drug: placebo — Subjects who were on placebo at Week 52 cannot continue in the extension treatment period
  Arms: placebo

SUMMARY:
The purpose of this study is to demonstrate efficacy of secukinumab at Week 12 based on PASI and IGA response rates versus placebo in subjects with moderate to severe chronic plaque-type psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Moderate and severe plaque-type psoriasis diagnosed for at least 6 months.
* Severity of psoriasis disease meeting all of the following three criteria:

Psoriasis Area and Severity Index (PASI) score of 12 or greater, Investigator's Global Assessment (IGA) score of 3 or greater, Total body surface area (BSA) affected of 10% or greater.

-Inadequate control by prior use of topical treatment, phototherapy and/or systemic therapy.

Exclusion criteria:

* Current forms of psoriasis other than chronic plaque-type psoriasis (for example, pustular, erythrodermic, guttate).
* Current drug-induced psoriasis.
* Previous use of secukinumab or any drug that targets IL-17 or IL-17 receptor.
* Significant medical problems such as uncontrolled hypertension, congestive heart failure or a condition that significantly immunocompromises the subject.
* Hematological abnormalities.
* History of an ongoing, chronic or recurrent infectious disease, or evidence of untreated tuberculosis.
* History of lymphoproliferative disease or history of malignancy of any organ system within the past 5 years.
* Pregnant or nursing (lactating) women. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2012-05-08 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (33):
- United States (18):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Glendale, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Newnan, Georgia
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Goodlettsville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Bryan, Texas
  - Novartis Investigative Site, Houston, Texas
- Canada (4):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, North Bay, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Québec
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (4):
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (5):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Osnabrück

REFERENCES:
- [Derived] Sticherling M, Nikkels AF, Hamza AM, Kwong P, Szepietowski JC, El Sayed M, Ghislain PD, Khotko AA, Patekar M, Ortmann CE, Forrer P, Papanastasiou P, Keefe D. Secukinumab in Pediatric Patients with Plaque Psoriasis: Pooled Safety Analysis from Two Phase 3 Randomized Clinical Trials. Am J Clin Dermatol. 2023 Sep;24(5):821-835. doi: 10.1007/s40257-023-00782-8. Epub 2023 Jun 21. PMID 37341961
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Houghton K, Patil D, Gomez B, Feldman SR. Correlation Between Change in Psoriasis Area and Severity Index and Dermatology Life Quality Index in Patients with Psoriasis: Pooled Analysis from Four Phase 3 Clinical Trials of Secukinumab. Dermatol Ther (Heidelb). 2021 Aug;11(4):1373-1384. doi: 10.1007/s13555-021-00564-2. Epub 2021 Jun 10. PMID 34110605
- [Derived] Menter A, Cather JC, Jarratt M, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab on Moderate-to-severe Plaque Psoriasis Affecting Different Body Regions: a Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):639-647. doi: 10.1007/s13555-016-0140-7. Epub 2016 Aug 30. PMID 27576559
- [Derived] Kircik L, Fowler J, Weiss J, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab for Moderate-to-Severe Head and Neck Psoriasis Over 52 Weeks: Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):627-638. doi: 10.1007/s13555-016-0139-0. Epub 2016 Aug 30. PMID 27573260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: "Study terminated by Sponsor" refers to the fact that - as per protocol - patients had to stop participating in the study in a given country where Secukinumab became available following approval.
Groups:
- AIN457 150 mg: Patients received one secukinumab 150 mg s.c. injection plus one placebo secukinumab s.c. injection at each dosing. In the open label phase only one 150 mg s.c. injection at each dosing
- AIN457 300 mg: Patients received two secukinumab 150 mg s.c. injections at each dosing
- Placebo - AIN457 150mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re- randomized to AIN457 150 mg for the remainder of the study
- Placebo - AIN457 300mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 300 mg for the remainder of the study
- Placebo: Patients received placebo secukinumab (2 s.c. injections) at each dosing
Period: Induction Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150mg | Placebo - AIN457 300mg | Placebo
Started | 59 | 59 | 0 | 0 | 59
Completed | 58 | 56 | 0 | 0 | 56
Not Completed | 1 | 3 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1
Not completed — Subject / guardian decision | 0 | 0 | 0 | 0 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150mg | Placebo - AIN457 300mg | Placebo
Started | 58 | 56 | 29 | 27 | 0
Completed | 48 | 52 | 25 | 25 | 0
Not Completed | 10 | 4 | 4 | 2 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Subject / guardian decision | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 6 | 1 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Period: Extension
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150mg | Placebo - AIN457 300mg | Placebo
Started | 46 | 51 | 23 | 23 | 0
Completed | 1 | 0 | 0 | 1 | 0
Not Completed | 45 | 51 | 23 | 22 | 0
Not completed — Adverse Event | 1 | 2 | 1 | 1 | 0
Not completed — Protocol deviation | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 6 | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0 | 0
Not completed — Study terminated by sponsor | 32 | 33 | 16 | 20 | 0
Not completed — Subject/guardian decision | 1 | 9 | 1 | 0 | 0
Not completed — Technical Problems | 1 | 0 | 0 | 1 | 0
Period: Follow-Up Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150mg | Placebo - AIN457 300mg | Placebo
Started | 36 | 31 | 19 | 18 | 0
Completed | 32 | 30 | 18 | 17 | 0
Not Completed | 4 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Subject / guardian decision | 3 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Total
Number analyzed (Participants) | 59 | 59 | 59 | 177
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46 (15.09) | 45.1 (12.57) | 46.5 (14.14) | 45.9 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 20 | 60
  Male | 40 | 38 | 39 | 117

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Secukinumab Compared to Placebo in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis at Week 12 Measure: PASI 75 (Psoriasis Area and Severity Index) Response.
Description: A 75% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI 75) is the current benchmark of primary endpoints for most clinical trials of psoriasis
Time Frame: 12 weeks
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 58 | 59
Percentage of participants | 69.5 | 75.9 | 0
Statistical Analysis 1: Comparison: AIN457 150 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: AIN457 300 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Primary Outcome: Efficacy of Secukinumab Compared to Placebo in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Measure:IGA (Investigator's Global Assessment) With a 0 or 1 Response at Week 12
Description: The IGA scale has been developed based on a previous version of the scale used in secukinumab phase II studies in collaboration with health authorities, in particular the FDA. The explanations/descriptions of the points on the scale have been improved to ensure appropriate differentiation between the points. The IGA used in this study is static, i.e. it refers exclusively to the subject's disease state at the time of the assessments, and does not attempt a comparison with any of the subject's previous disease states, whether at baseline or at a previous visit. IGA has a scale of 0-4 with the lower scores correlating to better performance. A score of 0= clear skin, 1= almost clear skin, 2=mild, 3=moderate,4=severe
Time Frame: 12 weeks
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 58 | 59
Percentage of Participants | 52.5 | 69 | 0
Statistical Analysis 1: Comparison: AIN457 150 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: AIN457 300 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Absolute Change From Baseline in Self Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 12
Description: The three domains of the POST SIAQ are feelings about injections, self-image, self-confidence, injection-site reactions, ease of use, and satisfaction with self-injection. The SIAQ items are scored on a semantic Likert-type scale where lower numbers indicate a worse experience. Domain scores range from 0 to 10. Subjects self-injecting at this visit completed this SIAQ questionnaire. The POST-SIAQ is taken after the injection at that visit.
Time Frame: Week 12
Population: Safety set: The safety set included all patients who took at least one dose of study treatment during the treatment period. Patients were analyzed according to treatment received
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 59 | 59
Score
  Feelings about injections | 1.07 (1.912) | 0.85 (1.685) | 0.57 (1.509)
  Self confidence | 1.10 (2.331) | 1.08 (2.197) | 1.26 (2.009)
  Satisfaction with self-injection | 1.64 (2.163) | 1.62 (2.667) | 1.32 (2.629)

4. Secondary Outcome: Absolute Change From Baseline in Self-Injection Assessment Questionnaire (SIAQ) Domain Scores at Week 48
Description: as for outcome 3
Time Frame: Baseline, week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Placebo-AIN457 150mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re- randomized to AIN457 150 mg for the remainder of the study
- Placebo-AIN457 300mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 300 mg for the remainder of the study
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo-AIN457 300mg
Number analyzed (Participants) | 58 | 56 | 29 | 27
Score
  Feelings about injections: number analyzed (Participants) | 45 | 52 | 25 | 24
  Feelings about injections | 0.93 (1.752) | 1.01 (2.103) | 0.63 (1.449) | 0.76 (1.321)
  Self-confidence: number analyzed (Participants) | 45 | 51 | 25 | 24
  Self-confidence | 1.63 (3.173) | 1.24 (2.400) | 0.97 (1.811) | 0.94 (1.521)
  Satisfaction, self-injection: number analyzed (Participants) | 43 | 50 | 25 | 23
  Satisfaction, self-injection | 1.92 (2.239) | 2.15 (2.673) | 1.90 (3.250) | 0.54 (1.840)

5. Secondary Outcome: Number of Subjects With Potential Use Related Hazards at Week 1
Description: To assess potential use-related hazards with the secukinumab PFS for the subject
Time Frame: Week 1
Population: as for outcome 3
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 59 | 59
Number of participants
  Needle stick in a critical area: number analyzed (Participants) | 58 | 57 | 59
  Needle stick in a critical area | 0 | 0 | 0
  Needle stick in non-critical area: number analyzed (Participants) | 58 | 57 | 59
  Needle stick in non-critical area | 0 | 0 | 1
  Any part of the device swallowed: number analyzed (Participants) | 58 | 57 | 59
  Any part of the device swallowed | 0 | 0 | 0
  Allergic reaction to device material: number analyzed (Participants) | 58 | 57 | 59
  Allergic reaction to device material | 0 | 0 | 0
  Pain due to bent needle: number analyzed (Participants) | 58 | 57 | 59
  Pain due to bent needle | 0 | 0 | 0
  Any breakage of the device: number analyzed (Participants) | 58 | 57 | 59
  Any breakage of the device | 0 | 0 | 0
  Swallowing of material debris observed: number analyzed (Participants) | 58 | 57 | 59
  Swallowing of material debris observed | 0 | 0 | 0
  Any other problem: number analyzed (Participants) | 58 | 57 | 59
  Any other problem | 1 | 0 | 0
  Less than full dose administered: number analyzed (Participants) | 58 | 57 | 59
  Less than full dose administered | 1 | 0 | 0

6. Secondary Outcome: Percentage of Subjects With Successful Self Administration of Study Drug at Week 1
Description: To assess the subject's ability to follow instructions for use with the secukinumab PFS
Time Frame: Week 1
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 58 | 57 | 59
Percentage of participants | 100 | 100 | 100

7. Secondary Outcome: Percent of Responders With Psoriasis Area and Severity Index (PASI) Equal to or Greater Than 50, PASI 75, PASI 90, PASI 100, (Induction) With Non-responder Imputation
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50, 75, 90 and 100 were defined as participants achieving ≥ 50%, 75%, 90% or 100% improvement from baseline.
Time Frame: Week 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 59 | 59
Percentage of participants
  Week 12 PASI 50 | 86.4 | 87.9 | 5.1
  Week 12 PASI 90 | 45.8 | 60.3 | 0
  Week 12 PASI 100 | 8.5 | 43.1 | 0

8. Secondary Outcome: Percent of Responders With Psoriasis Area and Severity Index (PASI) Equal to or Greater Than 50, PASI 75, PASI 90, PASI 100, (Maintenance; Observed Data)
Description: as for outcome 7
Time Frame: Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of participants
Groups:
- Placebo - AIN457 300 mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 300 mg for the remainder of the study
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 59 | 58 | 29 | 27
Percentage of participants
  Week 52 PASI 75 | 71.4 | 84.6 | 72.0 | 96.0
  Week 52 PASI 50 | 89.8 | 96.2 | 84.0 | 100.0
  Week 52 PASI 90 | 59.2 | 69.2 | 64.0 | 76.0
  Week 52 PASI 100 | 36.7 | 48.1 | 52.0 | 44.0

9. Secondary Outcome: Percent of Responders With Investigator's Global Assessment (IGA) Mod 2011 Score of 0 or 1, (Maintenance; Observed Data)
Description: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 59 | 59 | 29 | 27
Percentage of participants | 51 | 71.2 | 72 | 92

10. Secondary Outcome: Absolute Change From Baseline for PASI Score at Week 12, (Induction)
Description: PASI: Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head:01, arms:0.2 body:0.3 legs:0.4)
Time Frame: Week 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 59 | 59
Units on a scale | -16.33 (8.49) | -17.90 (8.74) | 0.50 (7.22)

11. Secondary Outcome: Absolute Change From Baseline for PASI Score Over Time up to Week 52, (Maintenance; Observed Data)
Description: as for outcome 10
Time Frame: Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 59 | 58 | 29 | 27
Units on a scale | -16.9 (8.27) | -18.7 (8.48) | -15.2 (5.38) | -20 (7.96)

12. Secondary Outcome: Number of Participants in Each Investigator's Global Assessment (IGA) Mod 2011 Category at Week 12, (Induction)
Description: The IGA mod 2011 category scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe
Time Frame: Week 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 58 | 59
Number of participants
  clear | 6 | 26 | 0
  almost clear | 26 | 17 | 0
  mild | 12 | 9 | 1
  moderate | 14 | 5 | 34
  severe | 1 | 1 | 24

13. Secondary Outcome: Percentage of Participants in Each Investigator's Global Assessment (IGA) Mod 2011 Category Over Time up to Week 52, (Maintenance; Observed Data)
Description: as for outcome 12
Time Frame: Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 59 | 59 | 29 | 27
Percentage of participants
  Clear | 36.7 | 48.1 | 52 | 44
  Almost clear | 14.3 | 23.1 | 20 | 48
  Mild | 18.4 | 19.2 | 4 | 4
  Moderate | 26.5 | 9.6 | 20 | 4
  Severe | 4.1 | 0 | 4 | 0

14. Secondary Outcome: Change From Baseline in EQ-5D at Week 12 (Induction)
Description: ED-5Q: Participant rated questionnaire to assess health related quality of life in terms of a single utility score. Five domains are assessed mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with three possible score: 1 indicates no problems, better state of health; 3 indicates worst state of health (example "confined to bed") A visual analog scale (VAS) assesses the health status from 0 (worst possible health state) to 100 (best possible health state)
Time Frame: Week 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 59 | 59 | 59
Units on a scale | 12.1 (24.03) | 11.2 (18.02) | 0.8 (16.12)

15. Secondary Outcome: Change From Baseline in EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D) Over Time up to Week 52, (Maintenance)
Description: as for outcome 14
Time Frame: Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo-AIN457 300mg
Number analyzed (Participants) | 57 | 57 | 29 | 26
Units on a scale | 11.4 (24.79) | 13.5 (15.69) | 12.2 (15.05) | 19.7 (17.16)

16. Secondary Outcome: Median Percentage Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score, (Induction)
Description: The DLQI is a quality of life measure used in the psoriatic The 10-item questionnaire has a score range of 0 (best) to 30 (worst) with higher scores indicating poor quality of life. The instrument contains six functional scales (i.e., symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment). Each item has 4 response categories, ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions. This result was reflected in the percentage change from baseline at Week 12, higher reductions (improvements) in DLQI scores (median treatment difference).
Time Frame: Baseline and week 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 56 | 53 | 54
Percent change | -78.6 [-85.9 to -67.5] | -85.0 [-90.9 to -77.7] | -16.7 [-25.3 to -3.0]

17. Secondary Outcome: Median Percentage Change From Baseline in Dermatology Life Quality Index (DLQI) Score Over Time up to Week 52, (Maintenance)
Description: as for outcome 16
Time Frame: Baseline and week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo-AIN457 300mg
Number analyzed (Participants) | 57 | 56 | 29 | 26
Percent change | -71.4 [-83.3 to -61.9] | -90.5 [-95.7 to -84.2] | -91.7 [-100 to -81.7] | -97.2 [-100 to -83.3]

18. Secondary Outcome: Percentage of Participants Achieving a DLQI Score of 0 or 1 at Week 12, (Induction)
Description: The DLQI is a quality of life measure used in the psoriatic The 10-item questionnaire has a score range of 0 (best) to 30 (worst) with higher scores indicating poor quality of life. The instrument contains six functional scales (i.e., symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment). Each item has 4 response categories, ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions
Time Frame: Week 12
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 57 | 53 | 54
Percentage of participants | 54.4 | 54.7 | 7.4

19. Secondary Outcome: Percentage of Participants Achieving a DLQI Score of 0 or 1 Over Time up to Week 52, (Maintenance)
Description: as for outcome 18
Time Frame: Week 52
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Number; unit: Percentage of participants
Groups:
- Placebo-AIN457 150 mg: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12, were re randomized to AIN457 150 mg for the remainder of the study
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150 mg | Placebo-AIN457 300mg
Number analyzed (Participants) | 28 | 35 | 18 | 20
Percentage of participants | 48.3 | 62.5 | 62.1 | 76.9

20. Secondary Outcome: Number of Responders With PASI Equal to or Greater Than 50, PASI 75, PASI 90, PASI 100 After Week 52
Description: as for outcome 7
Time Frame: Week 172
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned. Results after Week 172 and beyond cannot be interpreted meaningfully due to low number of evaluable patients at these visits.
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 59 | 59 | 29 | 27
Number of participants
  Week 172 PASI 75: number analyzed (Participants) | 27 | 32 | 13 | 19
  Week 172 PASI 75 | 26 | 25 | 9 | 17
  Week 172 PASI 50: number analyzed (Participants) | 27 | 32 | 13 | 19
  Week 172 PASI 50 | 27 | 32 | 12 | 18
  Week 172 PASI 90: number analyzed (Participants) | 27 | 32 | 13 | 19
  Week 172 PASI 90 | 14 | 21 | 9 | 11
  Week 172 PASI 100: number analyzed (Participants) | 27 | 32 | 13 | 19
  Week 172 PASI 100 | 6 | 16 | 6 | 7

21. Secondary Outcome: Absolute Change From Baseline for PASI Score After Week 52, (Observed Data)
Description: as for outcome 10
Time Frame: Week 172
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 27 | 32 | 13 | 19
Units on a scale | -18 (6.97) | -18.7 (8.36) | -14.7 (5.97) | -19.4 (9.02)

22. Secondary Outcome: Number of Participants in Each IGA Mod 2011 Category After Week 52 (Observed Data)
Description: The IGA mod 2011 is a static scale, i.e., it refers exclusively to the participant's disease state at the time of the assessments and does not attempt a comparison to any of the participant's previous disease states at prior visits. The score ranges from 0 (clear) to 4 (severe. The score 0 is clear, 1 is almost clear, 2 is mild, 3 is moderate, and 4 is severe
Time Frame: Week 172
Population: as for outcome 20
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 59 | 59 | 29 | 27
Number of participants
  Clear: number analyzed (Participants) | 27 | 32 | 13 | 19
  Clear | 7 | 15 | 7 | 7
  Almost clear: number analyzed (Participants) | 27 | 32 | 13 | 19
  Almost clear | 3 | 4 | 1 | 2
  Mild: number analyzed (Participants) | 27 | 32 | 13 | 19
  Mild | 16 | 6 | 3 | 6
  Moderate: number analyzed (Participants) | 27 | 32 | 13 | 19
  Moderate | 1 | 7 | 1 | 4
  Severe: number analyzed (Participants) | 27 | 32 | 13 | 19
  Severe | 0 | 0 | 1 | 0

23. Secondary Outcome: Number of Participants Developing Treatment Emergent Anti-secukinumab Antibodies, Immunogenicity
Description: The development of anti-secunimubab anti-bodies will decrease a participant's ability to respond to secukinumab treatment. The number of participants developing anti-secukinumab anti-bodies was measured from Baseline to 8 weeks after last treatment
Time Frame: Baseline and at Week 12, 24, 52, 100, 148, and 196, 204
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo-AIN457 150mg | Placebo-AIN457 300mg | Placebo
Number analyzed (Participants) | 59 | 59 | 29 | 27 | 3
Number of participants | 3 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Treatment until Last Patient Last Visit, approximately 4 years.
Description: AE additional description
Groups:
- Induction AIN457 150 mg: Patients received one secukinumab 150 mg s.c. injection plus one placebo secukinumab s.c. injection at each dosing
- Induction AIN457 300 mg: Patients received two secukinumab 150 mg s.c. injections at each dosing
- Induction Placebo: placebo secukinumab (2 s.c. injections) at each dosing
- Entire Any AIN457 150 mg: Includes all patients in the AIN457 150 mg and in the placebo- AIN457 150 mg treatment groups
- Entire Any AIN457 300 mg: Includes all patients in the AIN457 300 mg and in the placebo- AIN457 300 mg treatment groups
Arm/Group | Induction AIN457 150 mg | Induction AIN457 300 mg | Induction Placebo | Entire Any AIN457 150 mg | Entire Any AIN457 300 mg
Serious Adverse Events (participants affected / at risk) | 1/59 | 3/59 | 1/59 | 10/88 | 10/86
Other Adverse Events (participants affected / at risk) | 29/59 | 24/59 | 22/59 | 70/88 | 74/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction AIN457 150 mg (N=59) | Induction AIN457 300 mg (N=59) | Induction Placebo (N=59) | Entire Any AIN457 150 mg (N=88) | Entire Any AIN457 300 mg (N=86)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 0 | 0 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 1 | 0
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 1 | 0
SEPTIC VASCULITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
ADENOSQUAMOUS CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction AIN457 150 mg (N=59) | Induction AIN457 300 mg (N=59) | Induction Placebo (N=59) | Entire Any AIN457 150 mg (N=88) | Entire Any AIN457 300 mg (N=86)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 5 | 0
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 1 | 0 | 2 | 3
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 2 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 4
COLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 5 | 2
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 3 | 5 | 1 | 10 | 7
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 5
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 5
NAUSEA (Gastrointestinal disorders) | 0 | 3 | 1 | 4 | 5
TOOTHACHE (Gastrointestinal disorders) | 2 | 0 | 1 | 10 | 4
VOMITING (Gastrointestinal disorders) | 0 | 2 | 0 | 4 | 6
ASTHENIA (General disorders) | 2 | 0 | 0 | 4 | 1
FATIGUE (General disorders) | 0 | 0 | 1 | 0 | 2
INJECTION SITE OEDEMA (General disorders) | 0 | 0 | 0 | 2 | 0
INJECTION SITE PAIN (General disorders) | 1 | 0 | 1 | 2 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 2 | 2
OEDEMA PERIPHERAL (General disorders) | 1 | 1 | 0 | 2 | 1
PYREXIA (General disorders) | 2 | 2 | 2 | 6 | 3
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 0 | 3 | 5
ABSCESS ORAL (Infections and infestations) | 0 | 0 | 0 | 0 | 2
ACARODERMATITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2
BRONCHITIS (Infections and infestations) | 0 | 1 | 1 | 5 | 4
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2
CONJUNCTIVITIS (Infections and infestations) | 0 | 1 | 0 | 2 | 1
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 1
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 2
FOLLICULITIS (Infections and infestations) | 0 | 0 | 1 | 2 | 2
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 5 | 4
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 2 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 4 | 6
LABYRINTHITIS (Infections and infestations) | 0 | 0 | 0 | 3 | 1
NASOPHARYNGITIS (Infections and infestations) | 3 | 3 | 5 | 21 | 17
ORAL CANDIDIASIS (Infections and infestations) | 1 | 1 | 0 | 1 | 2
ORAL HERPES (Infections and infestations) | 0 | 1 | 0 | 0 | 5
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 1 | 2
OTITIS MEDIA BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 2 | 0
PERIODONTITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 2
PHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 3 | 4
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 3
RHINITIS (Infections and infestations) | 2 | 1 | 0 | 7 | 5
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 7 | 3
SKIN BACTERIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 2 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2
TINEA PEDIS (Infections and infestations) | 0 | 0 | 0 | 0 | 3
TONGUE FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2
TONSILLITIS (Infections and infestations) | 0 | 0 | 1 | 5 | 2
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 0 | 2 | 2
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 3 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 1 | 16 | 16
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 5 | 4
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 6 | 3
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 | 1 | 0 | 2 | 5
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 2
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 4
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 2 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 2 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 0 | 0 | 2 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 2
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 2
HEPATIC ENZYME INCREASED (Investigations) | 0 | 1 | 0 | 0 | 2
VITAMIN D DECREASED (Investigations) | 0 | 0 | 0 | 2 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 2
WEIGHT INCREASED (Investigations) | 0 | 1 | 0 | 0 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 1 | 5 | 2
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
HYPOSIDERAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 7 | 11
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 4 | 6
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 3
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 5 | 6
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
HEADACHE (Nervous system disorders) | 4 | 0 | 4 | 5 | 6
MIGRAINE (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
SCIATICA (Nervous system disorders) | 0 | 1 | 0 | 0 | 5
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
SYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 3 | 3
DEPRESSION (Psychiatric disorders) | 2 | 1 | 0 | 6 | 2
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 3 | 1
GLYCOSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 2
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 2 | 1 | 0 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 8 | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 5 | 10
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 2
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 3
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 5
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 3
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 6 | 3
URTICARIA PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
HAEMATOMA (Vascular disorders) | 0 | 1 | 0 | 0 | 3
HYPERTENSION (Vascular disorders) | 2 | 1 | 1 | 3 | 3

LIMITATIONS AND CAVEATS:
Since most patients were discontinued from study once secukinumab was commercially available in the respective countries, results beyond week 172 cannot be interpreted meaningfully.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial